CLINICAL TRIAL: NCT00005652
Title: Phase II Study of Rituximab in Patients With Immune Thrombocytopenic Purpura
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/15038; UAB-9866; UAB-BB-IND-8136; UAB-F990224001
Record Dates: First submitted 2000-05-02; First posted 2000-05-03 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2008-09

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic
Keywords: hematologic disorders; immune thrombocytopenic purpura; rare disease
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Hematologic Diseases; Rare Diseases | interventions — Rituximab

INTERVENTIONS:
Drug: rituximab

SUMMARY:
OBJECTIVES: I. Determine the response rate and response duration to rituximab in patients with immune thrombocytopenic purpura.

II. Evaluate the toxicity associated with this treatment regimen in these patients.

III. Evaluate the alteration in antiplatelet antibody with this treatment regimen in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive rituximab IV on days 1, 8, 15, and 22. Patients who achieve a clinical response lasting over 4 months may receive a second course of rituximab.

Patients are followed at 5, 6, 8, and 12 weeks, and then at 6 and 9 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Clinically confirmed immune thrombocytopenic purpura (ITP) Platelet count less than 75,000/mm3 on two occasions at least 1 week apart within past month

Normal to increased numbers of megakaryocytes on bone marrow examination within past 6 months

Failed prior steroid therapy (i.e., unable to achieve sustained platelet count greater than 75,000/mm3)

No drug associated ITP

No B cell malignancies

No evidence of disseminated intravascular coagulation (DIC)

--Prior/Concurrent Therapy--

Endocrine therapy: Concurrent steroids allowed as long as platelet count is less than 75,000/mm3 and dose is not changed within past 2 weeks or during study

Other:

* No other concurrent medical therapy for immune thrombocytopenia purpura (ITP)
* At least 2 weeks since prior therapy for ITP (except steroids)
* At least 4 weeks since prior cyclosporine

--Patient Characteristics--

Performance status: ECOG 0-2

Life expectancy: At least 6 months

Renal: Creatinine no greater than 2.0 mg/dL

Cardiovascular: No congestive heart failure or symptomatic coronary insufficiency

Other:

* No clinically significant bleeding (i.e., other than mild mucosal bleeding or petechiae)
* No sepsis or fever
* No active infection requiring therapy
* No active chronic viral infection
* HIV negative
* No other concurrent or prior malignancy within past 5 years except squamous or basal cell carcinoma of the skin or carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2000-12; Primary Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mansoor Noorali Saleh, Study Chair — University of Alabama at Birmingham
Locations (1):
- University of Alabama Comprehensive Cancer Center, Birmingham, Alabama, United States